CLINICAL TRIAL: NCT00003368
Title: Phase I Study of Irinotecan for Patients With Abnormal Liver or Renal Function or With Prior Pelvic Radiation Therapy
Brief Title: Irinotecan in Treating Patients With Solid Tumors or Lymphoma Who Have Abnormal Liver or Kidney Function or Who Have Received Radiation Therapy to the Pelvis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Purpose: Treatment
Other Study IDs: CDR0000066357; U10CA031946 (NIH); CLB-9863
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2006-07

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Irinotecan may be effective in treating patients with abnormal liver or kidney function or who have received radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of irinotecan in treating patients with solid tumors or lymphoma who have abnormal liver or kidney function or who have had previous radiation therapy to the pelvis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan in patients with solid tumors or lymphoma who have liver or renal dysfunction or have had prior pelvic radiation. II. Characterize the pharmacokinetics of irinotecan in these patients.

OUTLINE: This is a dose escalation study. Patients are stratified according to prior pelvic radiation therapy (yes vs no). Patients with no prior pelvic radiation are further stratified according to AST, bilirubin, and creatinine levels. Patients receive irinotecan IV over 90 minutes every 3 weeks for a total of 2 courses. After patients are reevaluated, treatment may continue in the absence of disease progression or unacceptable toxicity. Cohorts of 3 to 6 patients receive escalating doses of irinotecan. Dose escalation proceeds within each stratum until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose below that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 75 patients will be accrued for this study at a rate of 2-3 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid tumors or lymphoma refractory to standard therapy or for which no standard therapy exists Brain metastases allowed if following criteria met: Asymptomatic Received prior therapy for brain metastases Stable for at least 2 months No concurrent steroid therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic and Renal: Albumin at least 2.5 g/dL Prothrombin time less than 1.6 For patients without prior pelvic radiotherapy: AST at least 3 times upper limit of normal (ULN) OR Bilirubin 1.0 - 7.0 mg/dL with any AST OR Creatinine 1.6 - 5.0 mg/dL For patients with prior pelvic radiotherapy: AST less than 3 times ULN AND Bilirubin less than 1.0 mg/dL AND Creatinine less than 1.6 mg/dL Other: Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony stimulating factors Chemotherapy: At least 4 weeks since prior chemotherapy (at least 6 weeks since melphalan or mitomycin) At least 3 months since suramin No prior nitrosoureas or irinotecan Endocrine therapy: No concurrent steroids (except as antiemetic for chemotherapy) Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 4 weeks since major surgery Other: No concurrent medications known to affect hepatic or renal function (e.g., antiseizure medication or nonsteroidal antiinflammatory drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan P. Venook, MD, Study Chair — University of California, San Francisco
Locations (45):
- United States (45):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Venook AP, Enders Klein C, Fleming G, Hollis D, Leichman CG, Hohl R, Byrd J, Budman D, Villalona M, Marshall J, Rosner GL, Ramirez J, Kastrissios H, Ratain MJ. A phase I and pharmacokinetic study of irinotecan in patients with hepatic or renal dysfunction or with prior pelvic radiation: CALGB 9863. Ann Oncol. 2003 Dec;14(12):1783-90. doi: 10.1093/annonc/mdg493. PMID 14630685